CLINICAL TRIAL: NCT02652962
Title: A Randomized, Double-blind, Placebo-Controlled, 4-Period Study Assessing the Safety, Tolerability and Glycemic and Appetite Effects of Gelesis200 Using Two Different Timings of Administration in Overweight and Obese Subjects
Brief Title: Gelesis200 Safety and Tolerability Study and Effects on Glycemic and Appetite Parameters
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-200-001
Record Dates: First submitted 2015-12-18; First posted 2016-01-12 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Overweight Obese
MeSH Terms: interventions — maltodextrin; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Gelesis200 x 2, 10 min (Experimental): 3 x 0.70g Gelesis200 capsules administered 10 minutes before each of 2 meals (breakfast, lunch).
  Interventions: Device: Gelesis200
- Gelesis200 x 2, 30 min (Experimental): 3 x 0.70g Gelesis200 capsules administered 30 minutes before each of 2 meals (breakfast, lunch).
  Interventions: Device: Gelesis200
- Placebo x 2, 10 min (Placebo Comparator): 3 x Placebo capsules administered 10 minutes before each of 2 meals (breakfast, lunch).
  Interventions: Other: Placebo
- Placebo x 2, 30 min (Placebo Comparator): 3 x Placebo capsules administered 30 minutes before each of 2 meals (breakfast, lunch).
  Interventions: Other: Placebo
- Gelesis200 x 3, 10 min (Experimental): 3 x 0.70g Gelesis200 capsules administered 10 minutes before each of 3 meals (breakfast, lunch, dinner).
  Interventions: Device: Gelesis200
- Gelesis200 x 3, 30 min (Experimental): 3 x 0.70g Gelesis200 capsules administered 30 minutes before each of 2 meals (breakfast, lunch).
  Interventions: Device: Gelesis200
- Placebo x 3, 10 min (Placebo Comparator): 3 x Placebo capsules administered 10 minutes before each of 3 meals (breakfast, lunch, dinner).
  Interventions: Other: Placebo
- Placebo x 3, 30 min (Placebo Comparator): 3 x Placebo capsules administered 30 minutes before each of 3 meals (breakfast, lunch, dinner).
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Gelesis200 — 3 capsules each containing 0.70 g
  Arms: Gelesis200 x 2, 10 min; Gelesis200 x 2, 30 min; Gelesis200 x 3, 10 min; Gelesis200 x 3, 30 min
Other: Placebo — 3 capsules each containing 0.57 g of a mixture of microcrystalline cellulose and maltodextrin in a ratio of approximately 50 ± 10%
  Other Names: maltodextrin/microcrystalline cellulose
  Arms: Placebo x 2, 10 min; Placebo x 2, 30 min; Placebo x 3, 10 min; Placebo x 3, 30 min

SUMMARY:
The purpose of this study is to determine the safety and tolerability of Gelesis200.

DETAILED DESCRIPTION:
This is a cross-over within parallel design. Parallel groups will receive Gelesis200 either 2 times or 3 times in one day before meals. Within the parallel groups, subjects will cross-over to 4 arms: A) Gelesis200 10 min before meals, B) Gelesis200 30 min before meals, C) Placebo 10 min before meals, D) Placebo 30 min before meals. Postprandial glucose, insulin and subjective appetite ratings will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-smoker (no use of tobacco products within 6 months prior to screening), ≥ 22 and ≤ 65 years of age, with BMI ≥ 27.0 and < 35.0 kg/m2.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 12 weeks prior to administration. Subjects vomiting within 24 hours pre-administration will be carefully evaluated for upcoming illness/disease. Inclusion pre-administration is at the discretion of the Qualified Investigator.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease, including, but not limited to pancreatitis, hepatitis B or C, HIV, swallowing disorders, and gastroesophageal reflux disease (at least 1 episode per week).
   3. the absence of clinically significant history of gastric or peptic ulcer, small bowel resection (except if related to appendectomy), intestinal stricture (e.g., Crohn's disease), intestinal obstruction or high risk of intestinal obstruction including suspected small bowel adhesions.
   4. the absence of clinically significant history or known presence of esophageal anatomic abnormalities (e.g., webs, diverticuli, rings), gastroparesis, and malabsorption.
   5. the absence of history of gastric bypass, any other gastric surgery and intragastric balloon.
   6. the absence of history of angina, coronary bypass, and myocardial infarction within 6 months prior to administration.
   7. the absence of history of abdominal radiation treatment.
   8. the absence of history of cancer within the past 5 years, except adequately-treated localized basal cell skin cancer.
3. Capable of consent.
4. Fasting plasma glucose ≥ 90 and <126 mg/dL (equivalent to ≥ 5.0 and < 7.0 mmol/L) at screening.

Notwithstanding the lower limit of 90 mg/dL (equivalent to 5.0 mmol/L), subjects with higher fasting plasma glucose will be prioritized, and efforts will be made to include subjects with fasting plasma glucose ≥ 100 mg/dL (equivalent to ≥ 5.6 mmol/L) in both cohorts.

Exclusion criteria

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to carboxymethylcellulose, citric acid, modified cellulose, microcrystalline cellulose, maltodextrin, gelatin, titanium dioxide, or other related substances.
4. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.
5. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
6. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
8. Participation in a clinical trial involving the administration of an investigational or marketed drug or device within 30 days (90 days for biologics) prior to the first administration or concomitant participation in an investigational study involving no drug or device.
9. Use of medication other than topical products without significant systemic absorption:

   1. prescription medication within 30 days prior to the first administration;
   2. over-the-counter products including natural health products (e.g., food supplements and herbal supplements) within 7 days prior to the first administration, with the exception of the occasional use of acetaminophen (up to 2 g daily);
   3. a depot injection or an implant of any drug within 3 months prior to the first administration.
10. Donation of plasma within 7 days prior to the first administration. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first administration.
11. Hemoglobin < 140 g/L and hematocrit < 0.37 L/L at screening.
12. Glycosylated hemoglobin (HbA1c ≥ 6.5% which is equivalent to ≥ 48 mmol/mol).
13. Serum low-density lipoprotein cholesterol ≥ 190 mg/dL (≥ 4.93 mmol/L).
14. Serum triglycerides ≥ 500 mg/dL (≥ 5.65 mmol/L).
15. Anticipating surgical intervention during the study.

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of Gelesis200 administered two times per day 10 min before meals evaluated through the assessment of AEs, vital signs, clinical laboratory parameters, and physical examination | 24 hours post administration
  Treatment-emergent AEs will be tabulated by treatment and cohort. Changes from baseline values in vital signs and clinical laboratory parameters will be evaluated.
Safety/tolerability of Gelesis200 administered three times per day 10 min before meals evaluated through the assessment of AEs, vital signs, clinical laboratory parameters, and physical examination | 24 hours post administration
  Treatment-emergent AEs will be tabulated by treatment and cohort. Changes from baseline values in vital signs and clinical laboratory parameters will be evaluated.
Safety/tolerability of Gelesis200 administered two times per day 30 min before meals evaluated through the assessment of AEs, vital signs, clinical laboratory parameters, and physical examination | 24 hours post administration
  Treatment-emergent AEs will be tabulated by treatment and cohort. Changes from baseline values in vital signs and clinical laboratory parameters will be evaluated.
Safety/tolerability of Gelesis200 administered three times per day 30 min before meals evaluated through the assessment of AEs, vital signs, clinical laboratory parameters, and physical examination | 24 hours post administration
  Treatment-emergent AEs will be tabulated by treatment and cohort. Changes from baseline values in vital signs and clinical laboratory parameters will be evaluated.

OTHER OUTCOMES:
Postprandial plasma glucose: AUC | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial plasma glucose: Tmax | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial plasma glucose: Cmax | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial serum insulin: AUC | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial serum insulin: Tmax | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial serum insulin: Cmax | -30 to 210 min post meal (two meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch
Postprandial subjective appetite ratings using 100mm visual analog scales anchored at the 2 extremes: AUC | -30 to 210 min post meal (two or three meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch. The VAS comprise 6 questions about hunger, thirst, satiety, fullness, prospective eating and drinking. Each question is scored separately.
Postprandial subjective appetite ratings using 100mm visual analog scales anchored at the 2 extremes: Cmax | -30 to 210 min post meal (two or three meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch. The VAS comprise 6 questions about hunger, thirst, satiety, fullness, prospective eating and drinking. Each question is scored separately.
Postprandial subjective appetite ratings using 100mm visual analog scales anchored at the 2 extremes: Tmax | -30 to 210 min post meal (two or three meals)
  Blood samples collected at -30, -10, 0, 30, 60, 90, 120, 150, 180, and 210 minutes relative to the beginning of breakfast and lunch. The VAS comprise 6 questions about hunger, thirst, satiety, fullness, prospective eating and drinking. Each question is scored separately.

CONTACTS AND LOCATIONS:
Overall Officials: Audet, Principal Investigator — Quebec City, Quebec Canada
Locations (1):
- Québec, Quebec, Canada